CLINICAL TRIAL: NCT06917677
Title: Hormonal Balance in the Mobilization-Fatigue-Recovery Cycle: Dynamics of the Physiological and Psychological Response to Pre-Competitive Stress
Brief Title: Hormonal Balance in Stress, Fatigue, and Recovery: Dynamics of Pre-Competition Responses
Status: Completed | Type: Observational
Sponsor: Poznan University of Physical Education (Other)
Responsible Party: Sponsor
Other Study IDs: Rowers 2023a
Record Dates: First submitted 2025-04-01; First posted 2025-04-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2023-10

CONDITIONS: Healthy
Keywords: Athletes; Fatigue; Recovery; Anxiety
MeSH Terms: conditions — Fatigue; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Blood samples will be collected using two types of polyethylene tubes:
  1) 4.9 mL tubes containing dipotassium EDTA (EDTAK₂) as an anticoagulant for plasma-based analyses; 2) 9 mL tubes with a clotting activator for serum preparation.
  Samples will be processed, aliquoted, and stored at -80°C for subsequent hormonal and biochemical analyses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Rowers: A single group of national-level rowers performing a 2000-meter maximal effort test as part of a qualification process. All participants undergo the same protocol with repeated measurements before and after exercise.
  Interventions: Behavioral: 2000-meter maximal effort test on rowing ergometer

INTERVENTIONS:
Behavioral: 2000-meter maximal effort test on rowing ergometer — Participants will perform a 2000-meter maximal effort test on a Concept II rowing ergometer, aiming to complete the distance in the shortest possible time. The test simulates a competitive race and serves as a qualification trial. It will be conducted under medical supervision and is intended to induce a high level of physiological and psychological stress representative of elite competition.

SUMMARY:
This observational study investigates how elite athletes respond physiologically and psychologically to pre-competitive stress in the context of a high-stakes performance test. The study focuses on the dynamic changes in stress-related hormonal biomarkers and self-reported psychological states across three key phases: mobilization (pre-exercise anticipation), fatigue (immediate post-effort), and recovery (1 hour and 24 hours post-exercise). The performance test serves as part of a qualification process for national and international championship competitions, providing an ecologically valid model of competitive stress. Blood samples and validated psychological questionnaires are used to assess hormonal fluctuations and subjective stress responses at four time points.

The main question it aims to answer is:

How do key hormonal markers and self-reported psychological stress levels change across the mobilization-fatigue-recovery cycle surrounding a competitive performance?

DETAILED DESCRIPTION:
Elite athletes frequently experience intense psychological and physiological stress before and during high-stakes competitions. While a certain level of pre-competitive stress is necessary for optimal performance, excessive or poorly regulated stress can negatively affect both performance outcomes and recovery. The body's response to stress involves complex neuroendocrine mechanisms, including the activation of the hypothalamic-pituitary-adrenal (HPA) axis and the release of stress-related hormones and neuromodulators. These include cortisol, testosterone, dopamine, serotonin, β-endorphins, and endocannabinoids such as anandamide and 2-arachidonoylglycerol (2-AG).

This observational cohort study aims to explore the dynamic changes in both hormonal and psychological stress responses across four time points-before, immediately after, 1 hour after, and 24 hours after-a standardized, high-intensity rowing performance test. This test is part of the official national team selection process and simulates the psychological and physical demands of real-world competition, making it an ecologically valid model for investigating stress.

Participants are elite rowers (men and women) who are current members of the national team. The test represents a critical selection tool for major championship events (e.g., World and National Championships), creating a natural, high-pressure environment to study pre-competitive stress. All participants provide blood samples at four time points and complete validated psychological questionnaires (including CSAI-2 and SCAT) before the test.

The study's primary outcomes include blood concentrations of stress- and motivation-related hormones (cortisol, testosterone, dopamine, serotonin, β-endorphin, anandamide, 2-AG), and scores from standardized psychological stress inventories assessing cognitive anxiety, somatic anxiety, and self-confidence. These variables are evaluated across the mobilization-fatigue-recovery cycle to capture both immediate and delayed responses to competitive stress.

Secondary outcomes include anthropometric measurements (height, body weight, body mass index, body composition, and training history), which will be used to describe the participant cohort and assess potential moderating factors.

This study is novel in its scope and methodology, integrating a broad panel of biological stress markers with subjective psychological assessments across multiple time points. While previous research has focused primarily on cortisol in isolated pre- or post-competition measures, this study tracks dynamic, time-resolved changes across the full stress-recovery spectrum. Furthermore, the inclusion of dopamine, β-endorphins, and endocannabinoids represents a rare and innovative attempt to explore less-studied but potentially critical components of the athlete stress response.

This study will provide new insights into the mechanisms of resilience, adaptation, and recovery in elite sport by evaluating how hormonal and psychological indicators shift together or diverge. Findings may help coaches, sports psychologists, and medical professionals better monitor athlete well-being, identify signs of overreaching or maladaptive stress, and develop more personalized strategies for performance readiness and mental support.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-24 years
* Member of the national rowing team
* Actively participating in training and selection processes
* Medically cleared for high-intensity exercise by a team physician

Exclusion Criteria:

* Current injury or illness affecting physical performance
* Use of medications that may influence hormonal or psychological responses (e.g., corticosteroids, antidepressants, hormonal therapies)
* Diagnosed neurological, or endocrine disorders
* Refusal to provide blood samples or complete questionnaires

Ages: 19 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The Polish Youth Rowing Team
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-10-20 (Actual); Primary Completion 2023-10-25 (Actual); Study Completion 2023-12-02 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in cortisol level. | At rest (before the test), directly after the test, and after 1-hour and 24-hour recovery periods.
  Concentration of cortisol [ng/ml]. Immunoenzymatic assay method using a diagnostic ELISA Kit
Changes from baseline in testosterone level. | At rest (before the test), directly after the test, and after 1-hour and 24-hour recovery periods.
  Concentration of testosterone [ng/mL]. Immunoenzymatic assay method using a diagnostic ELISA Kit
Changes from baseline in serotonin level. | At rest (before the test), directly after the test, and after 1-hour and 24-hour recovery periods.
  Concentration of serotonin [ng/mL]. Immunoenzymatic assay method using a diagnostic ELISA Kit
Changes from baseline in dopamine level. | At rest (before the test), directly after the test, and after 1-hour and 24-hour recovery periods.
  Concentration of dopamine [ng/mL]. Immunoenzymatic assay method using a diagnostic ELISA Kit
Changes from baseline in beta-endorphin level. | At rest (before the test), directly after the test, and after 1-hour and 24-hour recovery periods.
  Concentration of beta-endorphin [ng/mL]. Immunoenzymatic assay method using a diagnostic ELISA Kit
Changes from baseline in anandamide level. | At rest (before the test), directly after the test, and after 1-hour and 24-hour recovery periods.
  Concentration of anandamide [ng/mL]. Immunoenzymatic assay method using a diagnostic ELISA Kit
Changes from baseline in 2-arachidonoyl glycerol level. | At rest (before the test), directly after the test, and after 1-hour and 24-hour recovery periods.
  Concentration of 2-arachidonoyl glycerol [ng/mL]. Immunoenzymatic assay method using a diagnostic ELISA Kit
Competitive Anxiety Profile Before Exercise Test Using SCAT Questionnaire | Before the 2000-meter exercise test (baseline, at rest)
  The Sport Competition Anxiety Test (SCAT) measures trait anxiety levels related to competitive situations in athletes. The SCAT questionnaire provides a score ranging from 10 to 30 points.
  Higher scores indicate higher levels of competitive anxiety, which is considered a worse outcome in terms of psychological readiness for competition.
  Lower scores suggest lower levels of trait anxiety and better psychological preparedness.
Cognitive, Somatic Anxiety, and Confidence Before and After Exercise Using CSAI-2R Questionnaire | Before the 2000-meter exercise test (baseline, at rest)
  The Competitive State Anxiety Inventory-2 Revised (CSAI-2R) measures the intensity of cognitive anxiety, somatic anxiety, and self-confidence in athletes before and after competitive performance. Each subscale of the CSAI-2R provides a score ranging from 9 to 36 points.
  For Cognitive Anxiety and Somatic Anxiety, higher scores indicate higher levels of anxiety, which are considered a worse outcome regarding psychological readiness.
  For Self-Confidence, higher scores indicate greater confidence, which is considered a better outcome.
Coping Strategies for Sport Stress Using CICS Questionnaire | Before the 2000-meter exercise test (baseline, at rest)
  The Coping Inventory for Competitive Sport (CICS) assesses athletes' coping strategies in response to competition-related stress. It measures task-oriented, distraction-oriented, and disengagement-oriented coping styles.
  Each subscale of the CICS (Task-Oriented Coping, Distraction-Oriented Coping, and Disengagement-Oriented Coping) provides a score ranging from 5 to 25 points.
  For Task-Oriented Coping, higher scores indicate more significant use of effective, adaptive coping strategies, which is considered a better outcome.
  For Distraction-Oriented Coping and Disengagement-Oriented Coping, higher scores indicate more significant use of less effective or maladaptive coping strategies, which is considered a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Skarpańska-Stejborn, Professor, Study Director — Poznań University of Physical Education, Faculty of Sport Sciences in Gorzów Wielkopolski, Poland;
Locations (1):
- Poznań University of Physical Education, Poznan, Greater Poland Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No